CLINICAL TRIAL: NCT04883619
Title: A Phase 2, Multicenter, Randomized, Double-Blind, Placebo-Controlled Study of Nipocalimab in Adult Participants With Active Lupus Nephritis
Brief Title: A Study of Nipocalimab in Adult Participants With Active Lupus Nephritis
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR109008; 80202135LUN2001 (Other: Janssen Research & Development, LLC); 2020-005568-79 (EudraCT Number)
Expanded Access: NCT05221619 (Temporarily not available)
Record Dates: First submitted 2021-05-11; First posted 2021-05-12 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Lupus Nephritis
MeSH Terms: conditions — Lupus Nephritis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Group 1: Placebo (Placebo Comparator): Participants will receive placebo intravenously (IV) every two weeks (q2w) from Week 0 through Week 50 along with standard-of-care treatment of mycophenolate mofetil (MMF) or mycophenolic acid (MPA) and glucocorticoid. Participants who will complete the assessments at Week 52 and have achieved complete renal response (CRR) may have the option to participate in the long-term extension (LTE) until unblinding of the study.
  Interventions: Other: Placebo; Drug: Standard-of-care treatment
- Group 2: Nipocalimab Dose 1 (Experimental): Participants will receive nipocalimab dose 1 IV q2w from Week 0 through Week 50 along with standard-of-care treatment of MMF or MPA and glucocorticoid. Participants who will complete the assessments at Week 52 and have achieved CRR may have the option to participate in the LTE of the study.
  Interventions: Drug: Nipocalimab; Drug: Standard-of-care treatment
- Group 3: Nipocalimab Dose 2 (Experimental): Participants will receive nipocalimab dose 2 IV q2w from Week 0 through Week 50 along with standard-of-care treatment of MMF or MPA and glucocorticoid. Participants who will complete the assessments at Week 52 and have achieved CRR may have the option to participate in the LTE of the study.
  Interventions: Drug: Nipocalimab; Drug: Standard-of-care treatment

INTERVENTIONS:
Other: Placebo — Placebo will be administered intravenously.
  Arms: Group 1: Placebo
Drug: Nipocalimab — Nipocalimab dose 1 and dose 2 will be administered intravenously.
  Other Names: JNJ-80202135; M281
  Arms: Group 2: Nipocalimab Dose 1; Group 3: Nipocalimab Dose 2
Drug: Standard-of-care treatment — Standard-of-care treatment including MMF or MPA and glucocorticoids will be administered intravenously through Week 52.

SUMMARY:
The purpose of this study is to evaluate the efficacy of nipocalimab versus placebo in participants with active Lupus Nephritis (LN).

DETAILED DESCRIPTION:
LN is a heterogeneous autoimmune disease that includes a broad spectrum of clinical forms, ranging from those with lesions confined to the skin (cutaneous lupus erythematosus [CLE]) to others that involve one or more vital internal organs (systemic lupus erythematosus [SLE]). Renal involvement due to SLE is termed LN. Nipocalimab (also referred to as JNJ-80202135 or M281) is a fully human aglycosylated immunoglobulin (Ig) G1 monoclonal antibody designed to selectively bind, saturate, and block the IgG binding site on the endogenous neonatal fragment crystallizable receptor (FcRn). By targeting the IgG binding site on FcRn, nipocalimab is expected to block the binding and, hence, recycling of IgG into circulation, resulting in a decrease in circulating IgG antibody levels, including pathogenic IgG autoantibodies and alloantibodies. The study will consist of a screening period (less than or equal to [<=] 8 Week), double-blind treatment period (52 Week), and a safety follow-up period (6 Week). Safety assessment will include adverse events (AEs), serious adverse events (SAEs), laboratory parameters (hematology and chemistry) and vital signs. The total duration of the main study is up to 66 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Kidney biopsy documentation of International Society of Nephrology (ISN)/Renal Pathology Society (RPS) proliferative nephritis: Class III or IV (with or without concomitant Class V) within the last 6 months prior to screening or performed during screening
* Urine Protein to Creatinine Ratio (UPCR) greater than or equal to (>=) 1.0 milligram/milligram (mg/mg) measured twice during screening
* Currently receiving prednisone equivalent dose of 1 milligram/kilogram/day (mg/kg/day) or less than or equal to (<=) 60 mg/day whichever is lower, or less. Must be receiving prednisone equivalent of 10 mg/day or more at screening and randomization. Treated for >= 6 weeks with stable dosing >= 2 weeks prior to first administration of study intervention
* If receiving angiotensin-converting enzyme (ACE) inhibitor/angiotensin II receptor blockers (ARB), a stable dose for at least 2 weeks prior to first administration of study intervention
* Is recommended to be up-to-date on all age-appropriate vaccinations prior to screening per routine local medical guidelines. For study participants who received locally-approved (and including emergency use-authorized) coronavirus disease 2019 (COVID-19) vaccines recently prior to study entry, follow applicable local vaccine labelling, guidelines, and standards-of-care for patients receiving immune-targeted therapy when determining an appropriate interval between vaccination and study enrolment

Exclusion Criteria:

* Comorbidities (other than Lupus Nephritis, example, asthma, chronic obstructive pulmonary disease) which have required 3 or more courses of systemic glucocorticoids within the previous 12 months
* Has other inflammatory diseases that might confound the evaluations of efficacy, including but not limited to rheumatoid arthritis (RA), psoriatic arthritis (PsA), RA/lupus overlap, psoriasis, Crohn's disease, or active Lyme disease
* Has received oral cyclophosphamide within 3 months or intravenous (IV) cyclophosphamide within 6 months prior to first administration of study intervention
* Has a history of latent or active granulomatous infection, including histoplasmosis or coccidioidomycosis, before screening
* COVID-19 infection: During the 6 weeks prior to baseline, have had any of the following (a) confirmed severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection (test positive), or (b) suspected SARS-CoV-2 infection (clinical features of COVID-19 without documented test results), or (c) close contact with a person with known or suspected SARS-CoV-2 infection

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2028-02-28 (Estimated); Study Completion 2028-02-28 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants Achieving Complete Renal Response (CRR) | Week 52
  Percentage of participants achieving complete renal response will be reported.

SECONDARY OUTCOMES:
Percentage of Participants Achieving CRR | Week 24
  Percentage of participants achieving CRR will be reported.
Percentage of Participants Achieving at Least 50 Percent (%) Decrease in Proteinuria from Baseline, Week 24 and Week 52 | Baseline, Week 24 and Week 52
  Percentage of participants achieving at least 50% decrease in proteinuria will be reported.
Percentage of Participants Achieving a Sustained Reduction in Steroid Dose Less Than or Equal to (<=)10 milligram (mg)/day of Prednisone or Equivalent | Week 16 to Week 52
  Percentage of participants achieving a sustained reduction in steroid dose <= 10 mg/day of prednisone or equivalent will be reported.
Percentage of Participants with Treatment-emergent Adverse Events (TEAEs) | Up to Week 66
  An adverse event (AE) is any untoward medical occurrence in a clinical study participant administered a pharmaceutical (investigational or non investigational) product. An AE does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. TEAEs are defined as AEs with onset or worsening on or after date of first dose of study treatment.
Percentage of Participants with Treatment-emergent Serious Adverse Events (TESAEs) | Up to Week 66
  A serious adverse event is any untoward medical occurrence that at any dose results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, is a suspected transmission of any infectious agent via a medicinal product. TESAEs are defined as SAEs with onset or worsening on or after date of first dose of study treatment.
Percentage of Participants with Treatment-emergent AEs Leading to Discontinuation of Study Intervention | Up to Week 52
  Percentage of participants with treatment-emergent AEs leading to discontinuation of study intervention will be reported.
Percentage of Participants with Treatment-emergent Adverse Events of Special Interests (AESIs) | Up to Week 58
  Percentage of participants with treatment-emergent AESIs will be reported.
Percentage of Participants with Change from Baseline in Laboratory Parameters Over Time | Up to week 58
  Percentage of participants with change from baseline in laboratory parameters (hematology and chemistry) will be reported.
Percentage of Participants with Change from Baseline in Vital Sign Parameters Over Time | Up to week 58
  Percentage of participants with change from baseline in vital sign parameters (temperature, pulse/heart rate, respiratory rate, and blood pressure) will be reported.
Serum Concentration of Nipocalimab Over Time | Up to Week 58
  Serum concentrations of nipocalimab over time in participants receiving active study intervention will be reported.
Number of Participants with Antibodies to Nipocalimab (Anti-Drug Antibodies [ADAs] and Neutralizing Antibodies [Nabs]) | Up to Week 58
  Number of participants with antibodies to nipocalimab (ADAs and Nabs) in participants receiving active study intervention will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency